CLINICAL TRIAL: NCT00151372
Title: Treatment Effectiveness in Depressed Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Treatment of Depressed Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: George S. Alexopoulos, M.D., Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201005319; R01HL071992-05 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2009-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Major Depression
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Adherence Intervention (Experimental): In the Treatment Adherence Intervention group, a study therapist regularly meets with subjects in order to identify obstacles to depression and chronic obstructive pulmonary disease treatment adherence and to help the participant overcome those obstacles.
  Interventions: Behavioral: Treatment Adherence Intervention
- Enhanced Care (Active Comparator): In the Enhanced Care group, physicians providing aftercare will be informed in writing of the patients' diagnosis but will receive no clinical instructions by the research team.
  Interventions: Behavioral: Enhanced Care

INTERVENTIONS:
Behavioral: Treatment Adherence Intervention — The care management intervention aims at facilitating adherence to a treatment algorithm based on the Agency for Health Care Policy and Research (AHCPR) guidelines. The investigators hypothesize that this intervention, in comparison to usual care, will increase the prescription of adequate antidepressant treatment by physicians, enhance treatment adherence by patients, and reduce depressive symptoms, suicide ideation, and disability.
  Arms: Treatment Adherence Intervention
Behavioral: Enhanced Care — For subjects in the Enhanced Care group, physicians providing aftercare will receive no clinical instructions by the research team, but will be informed in writing of the patients' diagnosis and will be provided with a copy of the Agency for Health Care Policy and Research (AHCPR) guidelines for the treatment of depression in primary care with an addendum updating the tables describing Selective Serotonin Reuptake Inhibitors (SSRI) side effect and dosage profiles. The investigators expect that these physicians will continue to base their practice on clinical judgment about how best to treat depression in chronic obstructive pulmonary disease patients.
  Arms: Enhanced Care

SUMMARY:
Approximately 20% of patients with chronic obstructive pulmonary disease (COPD) have major depression, a condition that contributes to suffering but also to poor treatment adherence leading to increased disability and morbidity. This study investigates the effectiveness of a care management intervention aimed at facilitating adherence to a treatment algorithm based on the Agency for Health Care Policy and Research (AHCPR) guidelines. The investigators hypothesize that this intervention, in comparison to usual care, will increase the prescription of adequate antidepressant treatment by physicians, enhance treatment adherence by patients, and reduce depressive symptoms, suicide ideation, and disability at a 28-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease by American Thoracic Society criteria
* Major depression by DSM-IV criteria
* 17-item Hamilton score >14
* English speaking

Exclusion Criteria:

* Inability to give informed consent
* MiniMental score <24
* Aphasia
* Nursing home placement after discharge

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2002-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George S Alexopoulos, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Helen Hayes Hospital, West Haverstraw, New York
  - Burke Rehabilitation Hospital, White Plains, New York
  - Weill Medical College of Cornell University, White Plains, New York

REFERENCES:
- [Derived] Solomonov N, Kerchner D, Bein O, Lee CE, Diaz JL, Ciarleglio A, Kim S, Sirey JA, Gunning FM, Raue PJ, Banerjee S, Arean PA, Alexopoulos GS. Precision Assignment to Psychosocial Interventions for Late-Life Depression: An Automated Treatment Decision Rule. JAMA Psychiatry. 2025 Nov 1;82(11):1075-1084. doi: 10.1001/jamapsychiatry.2025.2518. PMID 40960814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from the Inpatient Pulmonary Rehabilitation Units of the Burke Rehabilitation Hospital and Helen Hayes Rehabilitation Hospital. Recruitment began in March 2002 and ended in January 2008.
Groups:
- Treatment Adherence Intervention: In the Intervention group, a study therapist regularly meets with subjects in order to identify obstacles to depression and chronic obstructive pulmonary disease (COPD) treatment adherence and to help the participant overcome those obstacles.
Period: Overall Study
Arm/Group | Treatment Adherence Intervention | Enhanced Care
Started | 67 | 74
Completed | 38 | 45
Not Completed | 29 | 29
Not completed — Death | 12 | 11
Not completed — Lost to Follow-up | 5 | 5
Not completed — Too sick medically to continue | 5 | 6
Not completed — Withdrawal by Subject | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Adherence Intervention | Enhanced Care | Total
Number analyzed (Participants) | 67 | 74 | 141
Age Continuous [Mean (Standard Deviation); unit: years] | 71.24 (8.54) | 71.5 (8.0) | 71.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 51 | 93
  Male | 25 | 23 | 48
Region of Enrollment [Number; unit: participants]
  United States | 67 | 74 | 141

OUTCOME MEASURES:

1. Primary Outcome: Composite Antidepressant Score Scale (CAD)
Description: The Composite Antidepressant Score scale (CAD) describes the adequacy of an antidepressant's dosage. Scores range from 0-4 with 0, 1, and 2 signifying subthreshold or non-adequate therapeutic dosages while 3 and 4 signify a therapeutic/adequate dosage. The best value is 4 while the worst value is 0.
Time Frame: 28 Weeks
Population: Analysis was conducted on subjects actively participating in the study at the 28-week assessment. The number corresponds to "Completed" in the "Participant Flow" section.
Measure: Number; unit: Participants
Arm/Group | Treatment Adherence Intervention | Enhanced Care
Number analyzed (Participants) | 38 | 45
Participants
  Adequate Antidepressant Treatment | 29 (7.4) | 25 (9.3)
  Non-Adequate Antidepressant Treatment | 9 | 20

2. Secondary Outcome: Hamilton Depression Rating Scale
Description: The 17-item Hamilton Depression Rating Scale (HDRS) measures the severity of a depressive episode: the higher the score, the more severe the depression. The Best value is 0 and the Worst value is 52.
Time Frame: 28 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Treatment Adherence Intervention | Enhanced Care
Number analyzed (Participants) | 38 | 45
points on a scale | 9.2 (5.7) | 12.4 (6.0)

ADVERSE EVENTS:
Time Frame: 1 Year. The 14, 28, and 52 week assessments recorded any serious adverse event that had taken place since the previous assessment.
Description: This research study only tracked serious adverse events which included any incident which required that the subject seek medical attention (for example, specially scheduled physician's appointment, emergency room visit, and/or inpatient hospitalization) or death. We did not track adverse events: "0" in the adverse event section reflects this.
Arm/Group | Treatment Adherence Intervention | Enhanced Care
Serious Adverse Events (participants affected / at risk) | 38/67 | 46/74
Other Adverse Events (participants affected / at risk) | 0/67 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Adherence Intervention (N=67) | Enhanced Care (N=74)
Accidental Medication Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atrial Fibrilation (Cardiac disorders) | 0 (0) | 1 (1)
Back surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Brain cancer (General disorders) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2)
Cervical cancer (General disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Debility (General disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
Edema (Renal and urinary disorders) | 1 (1) | 2 (2)
Exacerbation of chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 25 (36) | 34 (38)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Heart attack (Cardiac disorders) | 1 (1) | 0 (0)
Heart surgery (Cardiac disorders) | 3 (4) | 0 (0)
High potassium levels (General disorders) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Inpatient psychiatric hospitalization (Psychiatric disorders) | 2 (2) | 1 (1)
Loss of consciousness/fainting (General disorders) | 1 (1) | 2 (2)
Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (5)
Renal Failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Staph infection (Infections and infestations) | 0 (0) | 3 (4)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Total knee replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Unknown case of death (General disorders) | 1 (1) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes